CLINICAL TRIAL: NCT04440137
Title: Controlling Early Childhood Caries and Terminating Bottle-feeding Habits Among Toddlers Using a Modified Oral Care Package: a Randomised Controlled Trial
Brief Title: Controlling ECC and Terminating Bottle-feeding Habits Among Toddlers Using a Modified Oral Care Package
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DRPG/08/19
Record Dates: First submitted 2020-05-31; First posted 2020-06-19 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Bottle Feeding; Dental Caries in Children
Keywords: Infant; Health promotion; Program development
MeSH Terms: conditions — Bottle Feeding

STUDY DESIGN:
Intervention Model Description: 1. Collection of Samples Randomization will be carried out.
  2. Research Briefing and Questionnaire Distribution Research briefing will be carried out and details of the study will be explained.
  3. Questionnaire Collection and Dental Examination at baseline
     1. After obtaining informed consent, questionnaires will be distributed.
     2. Caries experience of children will be recorded using ICDAS score. Caries experience also will be recorded in DMFT with cavitated and DMFT without cavitated.
     3. Intervention group will be provided with intervention brochure, kid toothbrush and toothpaste and a free-flow cup. Control group will receive brochure with standard of care info and kid toothbrush and toothpaste.
     4. An electronic form of OHP, will be given every 3 months to both group
     5. Dental check-up will be done every 6 months at the respective woman and child clinic.
     6. After a period of 1 year, the patient will be given a questionnaire again and dental check-up to compare any difference.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): Mother of children will receive a brochure with a standard of care info (with only essential information regarding the harmful effect of bottle feeding) and kid toothbrush and toothpaste (1000ppm of fluoride).
- Intervention group (Experimental): Mother of the children will be provided with intervention brochure (which include detailed information regarding the harmful effect of bottle feeding), kid toothbrush and toothpaste (1000ppm of fluoride) and a sippy cup.
  Interventions: Behavioral: Bottle-feeding cessation program

INTERVENTIONS:
Behavioral: Bottle-feeding cessation program — Specific brochure and proper oral hygiene education emphasizing on the benefit of stopping bottle-feeding given to subject
  Arms: Intervention group

SUMMARY:
This study will evaluate the effectiveness of oral health promotion in the prevention of ECC (early childhood caries) in bottle-fed children. Half of the patient will receive oral health promotion which emphasizing more on the benefit of stopping the bottle feeding habit, a free-flow cup and oral hygiene kit which include a toothbrush, toothpaste (1000ppm fluoride). The other half of the patient will receive standard of care oral hygiene promotion and oral hygiene kit which include a toothbrush, toothpaste (1000ppm fluoride)

DETAILED DESCRIPTION:
In Malaysia, even though there are decreasing trend in caries prevalence from a survey conduct in 1995 to 2015 (87.1% 1995, 76.2% 2005 and 71.3% 2015) [NOHPS 2015], yet the difference is just 15.8% in a period of 20 years. One of the factors which contribute to the development of ECC in children in prolonged bottle-feeding. Many literatures had mentioned association of bottle feeding and ECC however there are no controlled studies done on the effect of bottle feeding and ECC. Despite antenatal oral health promotion program done by Ministry of Health Malaysia and incorporation of oral hygiene education and oral hygiene instruction during dental visit, the prevalence of ECC remains high. This study will provide evidence regarding the effectiveness of oral health promotion in preventing early childhood caries by early termination of bottle feeding in toddlers.

ELIGIBILITY:
Inclusion Criteria:

* Malaysian citizen
* Child age 12 to 24 months old
* Child with bottle feeding habit (patients from Klinik Kesihatan Ibu & Anak (KKIA))
* Having at least 2 upper and 2 lower incisors at the time of recruitment
* A child is taken care of predominantly by their mother (housewife) or a single carer (maid/ grandmother)
* The parent who can read and write in Bahasa Melayu
* Full Term baby

Exclusion Criteria:

* Patient with medical problems
* Cleft lip or cleft palate or both
* Patient with a craniofacial anomaly

Ages: 1 Year to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-08-06 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
To identify changes in caries incidence | Baseline, 6 month, 12 month
  After the measurement of caries experience during the first visit, subject will be seen again in period of 6 month and 12 month to measure caries incidence on both group

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Haziq, Principal Investigator — Faculty Of Dentistry, University Of Malaya; Shani Ann Mani, Principal Investigator — Faculty Of Dentistry, University Of Malaya; Sharifah Wade'ah Wafa, Principal Investigator — Faculty Of Dentistry, University Of Malaya
Locations (1):
- Faculty Of Dentistry, University of Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No